CLINICAL TRIAL: NCT04002648
Title: Minimally Invasive or Conventional Edge-To-Edge Repair for Severe Mitral Regurgitation Due to Bileaflet Prolapse in Barlow's Disease: Does the Surgical Approach Have an Impact on the Long-term Results?
Status: Completed | Type: Observational
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Michele De Bonis, Principal Investigator, Ospedale San Raffaele
Other Study IDs: MICETE-BBL
Record Dates: First submitted 2019-06-27; First posted 2019-06-28 (Actual); Results first posted 2020-02-19 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Barlow's Disease; Prolapse; Mitral
MeSH Terms: conditions — Mitral Valve Prolapse | interventions — Sternotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MT-Right
  Interventions: Procedure: Right minithoracotomy
- Sternotomy
  Interventions: Procedure: Sternotomy

INTERVENTIONS:
Procedure: Right minithoracotomy — Incision of the right chest between 3rd and 4th or 4th and 5th intercostal space
  Groups: MT-Right
Procedure: Sternotomy — Longitudinal resection of the sternum
  Groups: Sternotomy

SUMMARY:
The study evaluates the long-term results of patients affected by bileaflet prolapse in Barlow's Disease, treated with edge-to-edge technique between 1997 and 2011.

ELIGIBILITY:
Inclusion Criteria:

Patients treated for bileaflet prolapse in Barlow's Disease between 1997 and 2011

Exclusion Criteria:

Age inferior to 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe MR due to the prolapse of both leaflets in the context of Barlow's disease submitted to EE repair via a video-assisted right minithoracotomy (minithoracotomy group) and patients with Barlow's disease treated with surgical mitral repair with the EE technique through a conventional median sternotomy (sternotomy group).
  The diagnosis of Barlow's disease was made during a preoperative transoesophageal echocardiographic (TEE) examination and confirmed by the surgeon's direct assessment of the valve. All patients had excessive leaflet tissue, annular dilatation and bileaflet prolapse. Cases with a forme fruste of Barlow's disease were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vahanian A, Alfieri O, Andreotti F, Antunes MJ, Baron-Esquivias G, Baumgartner H, Borger MA, Carrel TP, De Bonis M, Evangelista A, Falk V, Lung B, Lancellotti P, Pierard L, Price S, Schafers HJ, Schuler G, Stepinska J, Swedberg K, Takkenberg J, Von Oppell UO, Windecker S, Zamorano JL, Zembala M; ESC Committee for Practice Guidelines (CPG); Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC); European Association for Cardio-Thoracic Surgery (EACTS). Guidelines on the management of valvular heart disease (version 2012): the Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Eur J Cardiothorac Surg. 2012 Oct;42(4):S1-44. doi: 10.1093/ejcts/ezs455. Epub 2012 Aug 25. No abstract available. PMID 22922698

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MT-Right | Sternotomy
Started | 104 | 104
Completed | 102 | 104
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MT-Right | Sternotomy | Total
Number analyzed (Participants) | 104 | 104 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (8) | 51 (13) | 43.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 patients lost to follow-up
  Participants
    number analyzed (Participants) | 102 | 104 | 206
    Female | 68 | 38 | 106
    Male | 34 | 66 | 100
Region of Enrollment [Number; unit: participants] — Population: 2 patients lost to follow-up
  participants
    Italy: number analyzed (Participants) | 102 | 104 | 206
    Italy | 102 | 104 | 206

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Death
Description: The cumulative incidence function (CIF) of cardiac death at 12 years, with noncardiac death as a competing risk
Time Frame: 12 years
Measure: Number (95% Confidence Interval); unit: percentage of participants with event
Arm/Group | MT-Right | Sternotomy
Number analyzed (Participants) | 102 | 104
percentage of participants with event | 3.9 [0.6 to 13.3] | 3.8 [1.3 to 8.8]

2. Primary Outcome: Severe MR
Description: The cumulative incidence function (CIF) of recurrent mitral regurgitation (MR) >_ 3+, with death as the competing risk
Time Frame: 12 years
Measure: Number (95% Confidence Interval); unit: percentage of participants with event
Arm/Group | MT-Right | Sternotomy
Number analyzed (Participants) | 102 | 104
percentage of participants with event | 5.8 [1.8 to 13.4] | 11.4 [5.9 to 18.8]

ADVERSE EVENTS:
Arm/Group | MT-Right | Sternotomy
Serious Adverse Events (participants affected / at risk) | 11/102 | 10/104
Other Adverse Events (participants affected / at risk) | 0/102 | 0/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MT-Right (N=102) | Sternotomy (N=104)
Reoperation (Surgical and medical procedures) | 11 (11) | 10 (10)

LIMITATIONS AND CAVEATS:
Limitations due to retrospective design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes